CLINICAL TRIAL: NCT06548451
Title: Augmented Reality Assisted Lung Nodule Localization: a Multicentered, Prospective, Randomly Controlled, Non-inferiority Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xinghua Cheng, MD, Shanghai Chest Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ShanghaiChestAR_multicentered
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
Keywords: augmented reality; localization; sublobectomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR-guided group (Experimental): Application of augmented reality technique for percutaneous lung nodule localization.
  Interventions: Device: Augmented reality guided localization
- CT-guided group (No Intervention): Computerized tomography (CT) guided percutaneous lung nodule localization.

INTERVENTIONS:
Device: Augmented reality guided localization — In this study, AR was utilized to assist in the localization of pulmonary nodule during sublobectomy lung resection in patient to assess the accuracy of the technique.
  Arms: AR-guided group

SUMMARY:
With the popularization of CT screening, the detection rate of small lung nodules has greatly increased. Therefore, the clinical thoracoscopic lung nodule biopsy and sub-lobectomy for radical resection of lung cancer are greatly required. Accurate resection of lung nodule depends on precise localization of pulmonary nodules. However, preoperative CT-guided Hook- wire positioning under local anesthesia, which is the current primary localization method, requires high equipment and expense, and may cause physical and mental trauma to the patient. Augmented reality (AR) is an innovative technology that superimpose a virtual scene into the real environment by fusing images, videos, or computer-generated models with patients during surgical operations. It can visually display the anatomical structures of organs or lesions, which significantly improves surgical efficiency. This project intends to use AR technology to localize the solitary pulmonary nodule (SPN) before surgery, compared with CT-guided Hook-wire localization. Compared with the localization of SPNs under CT guidance, AR-assisted localization technology apparently is less time-consuming and can be performed immediately before surgery under general anesthesia, lessening pain, reduce costs of time and equipment, increase the success rate of sub-lobectomy, and improve the overall efficiency of surgical treatment of pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years inclusive;
2. No distant metastasis in preoperative clinical assessment;
3. The attending physician's assessment confirms the need for lung nodule localization in patients undergoing sublobar resection;
4. Target lung nodule diameter is no more than 2 cm;
5. The inner edge of the target nodule is at least 2 cm away from the pulmonary artery or pulmonary vein;
6. Non-pleural surface nodules;
7. Preoperative ECOG performance status score of 0/1;
8. Voluntarily participating in this study and signing an informed consent form.

Exclusion Criteria:

1. More than two lung nodules need to be removed at the same time.
2. The target node is located in the scapular region. Because percutaneous localization is obstructed by the scapula, percutaneous localization of pulmonary nodules is not suitable for such patients.
3. Patients with chronic pain issues or those who have been taking pain medications for an extended period.
4. Patients have uncontrollable mental illness and cannot make subjective assessment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of sublobar resection | 120 minutes
  The surgeon assesses whether effective lung sublobar resection has been achieved intraoperatively. Effective lung sublobar resection is defined as: (1) Completing planned sublobar resection in one session without the need for supplementary segmental or lobar resections; (2) Having a margin distance from the nodule of over 2 cm or at least 1 times the diameter of the nodule. If effective resection is not achieved, the proportion of supplementary segmental or lobar resections will be recorded.

SECONDARY OUTCOMES:
Operation duration | 30 minutes
  Since the start/end point of CT-guided pulmonary nodule localization may be arbitrary and there may be differences between different researchers, the program duration is derived from the CT scanning parameters and calculated as the length of time between the initial scan and the final scan. The augmented reality (AR) guided positioning time is automatically recorded by the system from the beginning of registration to the completion of positioning.
Interval time from localization to surgery | 60 minutes
  The time from completion of localization to the start of skin incision for surgery is calculated as the interval time from localization to surgery for both groups.
Complications related to nodule localization | 60 minutes
  1. CT-guided group: CT-guided localization is performed with the presence of research personnel or assistants to ensure compliance with the study protocol and to collect information on complications on-site. Occurrences of pneumothorax and pulmonary hemorrhage are immediately assessed after localization. Other rare complications such as vasovagal reactions and hemoptysis are also documented. After lung nodule localization, patients are taken to the anesthesia waiting area. During this time, nurses closely monitor the patients for worsening pneumothorax. Any occurrences of hemoptysis or other discomfort are meticulously recorded.
  2. AR-guided group: Due to the inability to assess pneumothorax and hemoptysis in AR-guided group, the anesthesiologist will be responsible for recording instances of airway bleeding and pneumothorax leading to decreased oxygen levels.
Radiation exposure dose | 30 minutes
  The dose length product (DLP) was used to quantify the total radiation received by patients during the localization of pulmonary nodules. In addition, after the scanning process, the DLP value is directly displayed on the screen of the CT scanner. In order to estimate the relative amount of radiation dose, the effective dose (ED) is also calculated according to the DLP value.
Dislodgement rate of the hookwire | 120 minutes
  The dislodgement of the hookwire is recorded by the operating surgeon or research assistant intraoperatively. Additionally, due to the impact of nodule depth on dislodgement rate, the distance between the lung nodule and the lung puncture point is also recorded.
Accuracy of nodule localization | 30 minutes
  The deviation between the hookwire and the target nodule center was evaluated. The deviation is expressed as vertical deviation, anteroposterior deviation and horizontal deviation in three dimensions. The total deviation of nodule localization is calculated as the square root of the sum of squares of each dimension.
Post-localization pain assessment | 40 days
  The post-localization pain assessment is conducted by the research assistant blindedly on the first day after surgery when the patient is fully awake. The assessment includes evaluating the patient's pain level during the localization process and at the localization site on the first day after surgery using the Numerical Rating Scale (NRS) for scoring. Additionally, pain assessment is repeated on the second day after surgery and again at 30 days after discharge (±7 days).
Post-localization trauma stress disorder assessment | 40 days
  The post-localization trauma stress disorder assessment is conducted by the research assistant in a blinded manner on the second day after surgery and at 30 days after discharge (±7 days). The Post-traumatic Stress Disorder Checklist - Civilian Version (PCL-C) is used to evaluates the psychological trauma experienced by patients due to the localization procedure.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - the people's second hospital Hefei, Hefei
  - Jiangyin Hospital of Traditional Chinese Medicine, Jiangyin
  - Jining No. 1 People's Hospital., Jining
  - Donghai County People's Hospital, Lianyungang
  - the First Hospital of Hebei Medical University, Shijia Zhuang
  - Zhangjiagang Hospital of Traditional Chinese Medicine,, Zhangjiagang